CLINICAL TRIAL: NCT02750852
Title: An Algorithm for Predicting Blood Loss and Transfusion Risk in Fast Track Total Hip Arthroplasty
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Azienda Ospedaliera Bolognini di Seriate Bergamo (Other)
Responsible Party: Principal Investigator, Riccardo Compagnoni, Medical doctor, Azienda Ospedaliera Bolognini di Seriate Bergamo
Other Study IDs: Blood algorithm
Record Dates: First submitted 2016-04-21; First posted 2016-04-26 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Total Hip Replacement; Blood Loss
MeSH Terms: conditions — Hemorrhage | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Analysis group: Create an algorithm to predict blood loss using patients data
  Interventions: Procedure: Total hip arthroplasty, blood loss analysis
- Control group: The algorithm was applied to analyze sensitivity and specificity
  Interventions: Procedure: Total hip arthroplasty, blood loss analysis

INTERVENTIONS:
Procedure: Total hip arthroplasty, blood loss analysis — Data analysis about blood loss in total hip replacement

SUMMARY:
Aim of these study is to create an algorithm, using data from patients that undergoing total hip arthroplasty, to predict blood loss after surgery and permit a safe domestic discharge.

DETAILED DESCRIPTION:
Two different cohorts of patients undergoing total hip arthroplasty will be analyzed to obtain data about hemoglobin trends. The first group will be used to obtain the algorithm, the second one to validate results of the first group, determining sensitivity and specificity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hip arthritis

Exclusion Criteria:

* ASA 4 - 5
* Active treatment with warfarin
* Coagulation disorders

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 124 patients, in two different cohorts, undergoing total hip arthroplasty.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2016-04; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Create an algorithm to predict blood loss after total hip arthroplasty | 3 months
  Data from the fist cohort of patients have been collected and analyzed to obtain an algorithm describing the trends of hemoglobin values after total hip arthroplasty. These algorithm was after applied to patients of a second cohort of consecutive patients undergoing total hip arthroplasty to determine specificity and sensitivity.

IPD SHARING:
Plan to Share IPD: No